CLINICAL TRIAL: NCT00975559
Title: The Relationship Between the Response to Mental Stress and Vascular Endothelial Function
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amir Lerman, M.D., Mayo Clinic
Other Study IDs: 1881-03
Record Dates: First submitted 2009-09-09; First posted 2009-09-11 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Endothelial Dysfunction; Apical Ballooning Syndrome; Myocardial Infarction
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Catecholomines
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal volunteers: Normal study volunteers with no prior history of coronary artery disease
- Apical Ballooning Syndrome: Women who have had a documented Apical Ballooning event as shown by coronary angiogram
- Coronary Endothelial Dysfunction: Patients who have been diagnosed with Endothelial Dysfunction via a coronary angiogram with acetylcholine challenge
- Myocardial Infarction: Women diagnosed with a Myocardial Infarction who subsequently had a Percutaneous Intervention

SUMMARY:
The aim of this study is to measure how different people respond to mental stress. The investigators will measure if there are differences in cardiovascular responses to mental stress among different groups of subjects. In one part of the study the investigators will compare the cardiovascular responses to mental stress between healthy women and healthy men. In another part of the study, the investigators will compare the cardiovascular responses to mental stress between women with apical ballooning syndrome and healthy post-menopausal women. The investigators hypothesize that healthy men will have an increased vascular response to and decreased endothelial function in response to to mental stress, compared to health women. Furthermore, the investigators hypothesize that women with apical ballooning syndrome will have an increased vascular response to and decreased endothelial function in response to mental stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be identified in one of the four groups outlined in "study population description."

Exclusion Criteria:

* Other co-morbidities that would make the testing not possible.
* Women who have had a mastectomy and would not have an arm that could be occluded during the reactive hyperemia portion of the Peripheral arterial tonometry testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Normal volunteers
  2. Apical Ballooning syndrome as proven during coronary angiogram
  3. Coronary Endothelial Dysfunction as proven during coronary angiogram
  4. Women who have had a Myocardial Infarction with subsequent Percutaneous Intervention
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2003-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States